CLINICAL TRIAL: NCT05624333
Title: Vegan Diets: the Short-term Effects on Daily Muscle Protein Synthesis Rates as Compared to Omnivorous Diets in Older Adults Assessed by D2O.
Acronym: VD2O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Rijksoverheid (Unknown); Maastricht University (Other)
Responsible Party: Principal Investigator, Lisette de Groot, Prof. Dr. Ir. L.C.P.G.M. (Lisette) de Groot, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: NL82653.028.22; NL9542 (Registry Identifier: Netherlands Trial Register); NL76916.028.21 (Other: METC Brabant)
Record Dates: First submitted 2022-11-08; First posted 2022-11-22 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Diet, Vegan; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VO group (Other): Vegan diet followed by Omnivorous diet
  Interventions: Other: Vegan diet (intervention); Other: Omnivorous diet (control)
- OV group (Other): Omnivorous diet followed by Vegan diet
  Interventions: Other: Vegan diet (intervention); Other: Omnivorous diet (control)

INTERVENTIONS:
Other: Vegan diet (intervention) — The intervention diet will be a fully controlled vegan diet that will be consumed for a duration of 10 days. No animal-based food products will be included in the diet.
Other: Omnivorous diet (control) — The control diet will be an a priori composed controlled omnivorous diet with a duration of 10 days. The omnivorous diet and the vegan diet will be isocaloric and isonitrogenous.

SUMMARY:
Consumers are increasingly encouraged to consume more plant-based foods and lower their consumption of foods from animal origin. However, the consequences of such a transition on muscle mass still remains to be explored. This is of particular importance in the older population, where sarcopenia is highly prevalent. The aim of this randomized controlled cross-over study is to investigate the short-term effect of a 10-day controlled vegan diet on daily muscle fractional synthesis rates in comparison to a 10-day controlled omnivorous diet in 35 community-dwelling older adults.

Participants will follow a fully controlled vegan diet, directly followed by a fully controlled omnivorous diet for 10 days, or vice versa. Researchers will compare the effect of the vegan diet to the effect of the omnivorous diet.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-79 years old;
* Community-dwelling;
* BMI 20-35 kg/m^2.

Exclusion Criteria:

* Following a vegetarian or vegan diet during the six months prior to the study;
* Following a diet that affects protein intake during the six months prior to the study;
* Participating in a structured exercise training program in the past three months;
* 5% or more body weight loss during three months before the start of the study;
* Being diagnosed with one of the following: diabetes; renal disease; neurological or neuromuscular disorders; serious cardiovascular diseases; cancer; chronic obstructive lung disease (COPD);
* Chronic use of medication that affects muscle function, e.g. corticosteroids, metformin, insulin;
* The use of the following medicines: acenocoumarol (sintrom); phenprocoumon (marcoumar); dabigatran (pradaxa); apixaban (eliquis); rivaroxaban (xarelto); clopidogrel (plavix); combination of acetylsalicylic acid or carbasalate calcium (ascal) with dipyridamole.
* Allergic or intolerant to any product included in the diets;
* Not willing to stop nutritional supplements, with the exception of supplements on medical advice, and vitamin D;
* Not willing or afraid to give blood or undergo a muscle biopsy during the study;
* Unwilling to eat a vegan and an omnivorous diet for ten days each;
* Currently a research participant in another trial or participated in a clinical trial during three months before the start of the measurement period;
* Not being able to understand Dutch;
* Not having a general physician.

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Muscle Protein Synthesis (MPS) | 10 days
  MPS, expressed as daily fractional synthesis rates (FSR, %/day), will be assessed using a deuterium oxide protocol. Daily FSR will be calculated using the 2^H-alanine enrichment in plasma and the mixed muscle-bound 2^H-alanine enrichment.

SECONDARY OUTCOMES:
Appetite | Measured daily for 10 days during each diet
  Appetite will be assessed using visual analogue scales (VAS; Min 0 mm - max 100 mm) before and after the warm meal. Five VAS-scales regarding hunger, fullness, satiation, desire to eat and prospective food consumption will be used to assess appetite.
Change in fasting plasma glucose | Change after 10 days of following each diet
  Fasting plasma glucose levels
Change in fasting plasma insulin | Change after 10 days of following each diet
  Fasting plasma insulin levels
Change in fasting plasma lipid profile | Change after 10 days of following each diet
  Triglycerides, high-density lipoprotein-cholesterol, low-density lipoprotein cholesterol, total cholesterol
Change in blood pressure | Change after 10 days of following each diet
  Fasting systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Lisette de Groot, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University and Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Domic J, Pinckaers PJ, Grootswagers P, Siebelink E, Gerdessen JC, van Loon LJ, de Groot LC. A Well-Balanced Vegan Diet Does not Compromise Daily Mixed Muscle Protein Synthesis Rates when Compared with an Omnivorous Diet in Active Older Adults: A Randomized Controlled Cross-Over Trial. J Nutr. 2025 Apr;155(4):1141-1150. doi: 10.1016/j.tjnut.2024.12.019. Epub 2024 Dec 26. PMID 39732437